CLINICAL TRIAL: NCT00564941
Title: Evaluating the Efficacy of Deferasirox in Transfusion Dependent Chronic Anaemias (Myelodysplastic Syndrome, Beta-thalassaemia Patients) With Chronic Iron Overload
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670AHU02
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Myelodysplastic Syndromes; Beta-Thalassemia
Keywords: Myelodysplastic Syndromes; beta-Thalassemia; Iron Overload; Iron Chelating Agents; deferasirox
MeSH Terms: conditions — Myelodysplastic Syndromes; beta-Thalassemia; Iron Overload | interventions — Deferasirox

ARMS (1):
- Deferasirox (Experimental)
  Interventions: Drug: deferasirox

INTERVENTIONS:
Drug: deferasirox
  Other Names: ICL670

SUMMARY:
This study will evaluate the safety and efficacy of deferasirox in transfusion dependent Myelodysplastic Syndrome, Beta-thalassaemia major patients with chronic iron overload

ELIGIBILITY:
Inclusion criteria:

* In- or outpatients with myelodysplasia / with risk of low or intermedier-1 according to the International Prognostic Scoring System (IPSS) confirmed by bone marrow evaluation within 3 month/ or beta thalassaemia major patients, who have chronic iron overload, as a consequence of frequent blood transfusion
* Serum ferritin> 1800 µg/L
* Age: 18-80 years
* men and women
* Chronic iron overload caused by at least 30 units and maximum 100 units of blood of packed red blood cells
* Deferoxamin therapy is contraindicated or inadequate or unable to use in the recommended dose due to intolerability or other reason
* Eastern Cooperative Oncology Group (ECOG) performance status score between 0-2
* written informed consent

Exclusion criteria:

* beta thalassaemia minor,
* haemosiderosis caused by other than chronic transfusional iron overload,
* patients with impaired renal function (Creatinin clearance< 60 ml/ min),
* pregnancy,
* lactation,
* patient of childbearing potential unwilling to use contraceptive precautions
* known hypersensitivity to deferasirox or any ingredients,
* impaired hepatic function (SGOT,SGPT 5x above UNL).
* Patients severely ill due to underlying disease progression or other severe concomitant disease.
* Patients with poor prognosis of karyotype
* patients with malabsorption caused by inflammatory bowel disease, gastrectomy, pancreatitis or other medical condition
* History of nephrotic syndrome
* Significant proteinuria
* Patients with a previous history of clinically relevant ocular toxicity related to iron chelation
* Patients with positive test to HIV

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Estimated)
Dates: Start 2007-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
This study will evaluate the safety and efficacy of deferasirox in transfusion dependent Myelodysplastic Syndrome, Beta-thalassaemia major patients with chronic iron overload | monthly during the therapy and at the end of the treatment (aftr 9 months therapy)

SECONDARY OUTCOMES:
patient's compliance during the study assessed by the number of the unused tablets returned by the patient safety assessed by patient laboratory data, adverse events, serious adverse events | during the treatment (9 months)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged